CLINICAL TRIAL: NCT04777721
Title: A Clinical Challenge Study to Evaluate Controlled Human Infection With BCG Administered by the Aerosol Inhaled Route in Historically BCG-vaccinated Healthy Adult Volunteers
Brief Title: Aerosol BCG Challenge Study in Historically BCG-vaccinated Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TB044
Record Dates: First submitted 2020-09-18; First posted 2021-03-02 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; BCG; Human challenge; Aerosol BCG challenge
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: This is a phase I dose-escalation clinical challenge study in historically BCG-vaccinated healthy adult volunteers in which BCG will be administered via the aerosol inhaled route.
  There will be four study groups with three volunteers in each group. Volunteers will be sequentially enrolled into each group in turn based on their availability. The first volunteer in each group will be challenged at least 1 hour apart from any subsequent volunteers. There will be a review of safety data at least 7 days after challenge of all volunteers within each dose group. This safety review will be performed by the Safety Monitoring Committee (SMC). Dose escalation into the next group will only occur if there are no safety concerns. Safety review will include assessment of symptom diary card, safety bloods and lung function results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: 1 x 10^4 cfu aerosol inhaled BCG (Experimental): 3 historically BCG-vaccinated volunteers will receive 1 x 10^4 cfu aerosol inhaled BCG. All Group 1 volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish
- Group 2: 1 x 10^5 cfu aerosol inhaled BCG (Experimental): 3 historically BCG-vaccinated volunteers will receive 1 x 10^5 cfu aerosol inhaled BCG. All Group 2 volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish
- Group 3: 1 x 10^6 cfu aerosol inhaled BCG (Experimental): 3 historically BCG-vaccinated volunteers will receive 1 x 10^6 cfu aerosol inhaled BCG. All Group 3 volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish
- Group 4: 1 x 10^7 cfu aerosol inhaled BCG (Experimental): 3 historically BCG-vaccinated volunteers will receive 1 x 10^7 cfu aerosol inhaled BCG. All Group 3 volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish

INTERVENTIONS:
Biological: BCG Danish — BCG Danish 1331 is on the WHO list of pre-qualified vaccines and has a well-defined side effect profile. BCG is licensed for delivery via the intradermal route. It is not licensed for delivery via the aerosol route.

SUMMARY:
The purpose of this study is to evaluate the human clinical response to BCG challenge in historically BCG-vaccinated healthy adult volunteers. It will involve 12 participants in a controlled dose escalation. Bronchoscopies will be performed 14 days post-challenge to measure BCG recovered from bronchial samples. Blood tests will be taken to look at potential immunological markers of immunity.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains one of the deadliest infectious disease killers worldwide. Key research priorities include the development of an effective vaccine.

Currently, the only licensed vaccine against TB is the BCG (Bacille Calmette-Guérin). This works well against TB in childhood but is often ineffective in adults. Developing a new TB vaccine is difficult, as it is hard to determine which will be effective. In other diseases, e.g. influenza or malaria, it is possible to experimentally-infect volunteers with the disease to see if the proposed vaccine is effective. This is called a "controlled human challenge or infection model" and is possible in easily treatable or self-limiting diseases. This is not possible with TB, where treatments may be harmful and complex. Using a related but less infectious bacterium is a feasible alternative.

The BCG is a live attenuated (weakened) strain of the bacteria that causes TB in cattle. The BCG bacteria do not cause disease in healthy individuals. As the BCG and TB bacteria are similar, a challenge model using the BCG as an infectious agent to mimic TB infection is being developed.

Mycobacterium tuberculosis, the bacterium that causes TB, infects people by inhalation into the lungs. Therefore, inhaled BCG more closely imitates TB infection than an injection. A previous (TB041) and current study (TB043) in this group use aerosol inhaled BCG in volunteers who have not received the standard BCG vaccination before.

The purpose of this study is to evaluate the human clinical response to BCG challenge in historically BCG-vaccinated healthy adult volunteers. It will involve 12 participants in a controlled dose escalation. Bronchoscopies will be performed 14 days post-challenge to measure BCG recovered from bronchial samples. Blood tests will be taken to look at potential immunological markers of immunity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-50 years
* Previously vaccinated with the BCG (at least 6 months prior to enrolment, as evidenced by a visible scar or documentation in medical or occupational health records)
* Resident in or near Oxford for the duration of the study period
* Provide written informed consent
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner (or review summary care record, if available)
* Allow the investigator to register volunteer details with a confidential database (The Over-volunteering Protection Service) to prevent concurrent entry into clinical studies/trials
* Agreement to refrain from blood donation during the course of the study
* For women of child-bearing potential only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening, challenge and bronchoscopy
* Able and willing (in the investigator's opinion) to comply with all study requirements
* No clinically relevant findings in medical history or on physical examination
* Screening IGRA negative
* Willing to be tested for evidence of SARS-CoV-2 infection and to allow public health notification of the results

Exclusion Criteria:

* Any clinically significant respiratory disease, including asthma
* Current smoker (defined as any smoking including e-cigarettes in the last 3 months)
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study agent, any essential study procedure, sedative drugs, or any local or general anaesthetic agents
* Clinically significant history of skin disorder, allergy, atopy, cancer (except BCC of the skin or CIS of the cervix), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* Any autoimmune conditions or immunodeficiency (including HIV)
* Previous diagnosis or treatment for TB disease or latent TB infections
* Clinical, radiological, or laboratory evidence of current active TB disease or latent TB infection
* Previous receipt of any investigational TB vaccine
* Positive HBsAg, HCV or HIV antibodies
* Concurrent use of oral, inhaled or systemic steroid medication or use for more than 14 days within the last 6 months (steroids used as a cream or ointment are permissible), or the use of other immunosuppressive agents concurrently or for more than 14 days within the last 6 months
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned study challenge date
* Current use of any medication or other drug taken through the nasal or inhaled route including cocaine or other recreational drugs
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Pregnancy, lactation or intention to become pregnant during study period
* Previously resident for more than 12 months concurrently in a tropical climate where significant non-tuberculous mycobacterial exposure is likely
* Shares a household with someone with clinically significant immunodeficiency (either from infection or medication) who is deemed to be at risk of developing disseminated BCG infection if exposed to BCG
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Clinically significant abnormality on screening chest radiograph
* Clinically significant abnormality of lung function testing
* Any clinically significant abnormality of screening blood or urine tests
* Laboratory confirmed (PCR or antibody) SARS-Cov-2 infection, evidence of viral pneumonitis on chest radiograph or a high clinical suspicion of COVID-19 disease in the 3 months preceding enrolment.
* A body mass index (BMI) of <18.5 or >45
* Any other significant disease, disorder, or finding, which, in the opinion of the investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the study or impair interpretation of the study data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Professor, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Fredsgaard-Jones T, Harris SA, Morrison H, Ateere A, Nassanga B, Ramon RL, Mitton C, Fletcher E, Decker J, Preston-Jones H, Jackson S, Mawer A, Satti I, Barer M, Hinks T, Bettinson H, McShane H. A dose escalation study to evaluate the safety of an aerosol BCG infection in previously BCG-vaccinated healthy human UK adults. Front Immunol. 2024 Nov 14;15:1427371. doi: 10.3389/fimmu.2024.1427371. eCollection 2024. PMID 39611145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: 1 x 10^4 Cfu Aerosol Inhaled BCG | Group 2: 1 x 10^5 Cfu Aerosol Inhaled BCG | Group 3: 1 x 10^6 Cfu Aerosol Inhaled BCG | Group 4: 1 x 10^7 Cfu Aerosol Inhaled BCG
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 1 x 10^4 Cfu Aerosol Inhaled BCG | Group 2: 1 x 10^5 Cfu Aerosol Inhaled BCG | Group 3: 1 x 10^6 Cfu Aerosol Inhaled BCG | Group 4: 1 x 10^7 Cfu Aerosol Inhaled BCG | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 1 | 1 | 1 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: To Quantify BCG Recoverable From Bronchial Sample
Description: Quantification of BCG culture by mycobacterial growth indicator tube (PCR quantification and DNA strip assay speciation as required)
Time Frame: Day 14
Measure: Number; unit: Volunteers with detectable BCG
Arm/Group | Group 1: 1 x 10^4 Cfu Aerosol Inhaled BCG | Group 2: 1 x 10^5 Cfu Aerosol Inhaled BCG | Group 3: 1 x 10^6 Cfu Aerosol Inhaled BCG | Group 4: 1 x 10^7 Cfu Aerosol Inhaled BCG
Number analyzed (Participants) | 3 | 3 | 3 | 3
Volunteers with detectable BCG | 0 | 0 | 0 | 0

2. Secondary Outcome: Adverse Events
Description: Evaluation of the human clinical response to BCG challenge via collection of data on adverse events at each visit, via diary cards and lung function test results.
Time Frame: Up to day 168
Measure: Number; unit: Number of participants reporting events
Arm/Group | Group 1: 1 x 10^4 Cfu Aerosol Inhaled BCG | Group 2: 1 x 10^5 Cfu Aerosol Inhaled BCG | Group 3: 1 x 10^6 Cfu Aerosol Inhaled BCG | Group 4: 1 x 10^7 Cfu Aerosol Inhaled BCG
Number analyzed (Participants) | 3 | 3 | 3 | 3
Number of participants reporting events | 3 | 1 | 3 | 3

3. Other Pre Specified Outcome: Identify Laboratory Markers of Immune Response That Correlate With the Levels of BCG Recovered From Bronchial and Other Samples.
Description: Laboratory markers of innate and adaptive immunity, determined by ex-vivo ELISpot
Time Frame: Up to day 168
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Identify Laboratory Markers of Immune Response That Correlate With the Levels of BCG Recovered From Bronchial Samples.
Description: Laboratory markers of innate and adaptive immunity, determined by ELISA
Time Frame: Up to day 168
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Identify Laboratory Markers of Immune Response That Correlate With the Levels of BCG Recovered From Bronchial Samples.
Description: Laboratory markers of innate and adaptive immunity, determined by RNA sequence analysis
Time Frame: Up to day 168
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Identify Laboratory Markers of Immune Response That Correlate With the Levels of BCG Recovered From Bronchial Samples.
Description: Laboratory markers of innate and adaptive immunity, determined by intracellular cytokine staining of blood and bronchial samples
Time Frame: Up to day 168
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Identify Laboratory Markers of Immune Response That Correlate With the Levels of BCG Recovered From Bronchial Samples.
Description: Laboratory markers of innate and adaptive immunity, determined by BCG cfu counts and or molecular diagnostics on induced sputum
Time Frame: Up to day 168
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Identify Laboratory Markers of Immune Response That Correlate With the Levels of BCG Recovered From Bronchial Samples.
Description: Laboratory markers of innate and adaptive immunity, determined by matrix from adapted mask collection
Time Frame: Up to day 168
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs reported within 72 hours of challenge
Arm/Group | Group 1: 1 x 10^4 Cfu Aerosol Inhaled BCG | Group 2: 1 x 10^5 Cfu Aerosol Inhaled BCG | Group 3: 1 x 10^6 Cfu Aerosol Inhaled BCG | Group 4: 1 x 10^7 Cfu Aerosol Inhaled BCG
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 1 x 10^4 Cfu Aerosol Inhaled BCG (N=3) | Group 2: 1 x 10^5 Cfu Aerosol Inhaled BCG (N=3) | Group 3: 1 x 10^6 Cfu Aerosol Inhaled BCG (N=3) | Group 4: 1 x 10^7 Cfu Aerosol Inhaled BCG (N=3)
Night Sweat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shivers (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temperature (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Feverishness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cough (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Sore throat (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tickly throat (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough phlegm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough Blood (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT04777721/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT04777721/ICF_001.pdf